CLINICAL TRIAL: NCT04434521
Title: Comparison of Different Refraction Measurements in Adults
Acronym: REFRACT
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PBMD04; 2020-A00259-30 (Other: IDRCB)
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Vision Loss Night
MeSH Terms: conditions — Vitamin A Deficiency | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire about habits in terms of near vision activities
Other: Eye examination — The eye examination involves the following measurements:
  * Distant vision phoria with Thorington method
  * Close vision with Thorington method
  * Objective eye-to-eye refraction with self-refractometer
  * Binocular objective refraction with autorefractometer
  * Monocular/biocular/binocular refraction with Nidek TS610
  * SiView automatic refraction
  * Humphriss binocular refraction
  * MOU Binocular refraction

SUMMARY:
The combatant is likely to carry out missions any time, any place, day or night. The very strong degradation of natural vision performance in these conditions justifies the use of visual replacement means, based on optronic sensors whose sensitivity is more adapted to these luminous environments than that of the human eye.

The duration and repetition of missions carried out with night vision sensors lead to visual complaints from users.

The literature on night vision binoculars adjustment states that a binocular adjustment of the equipment provides more convex settings. The latter would then limit the strain on the accommodative component, which is one of the possible sources of operator visual fatigue. In order to allow a more appropriate adjustment, it is proposed to rely on a measurement of the refraction (optical defect of the eye) of each operator. Like binocular adjustments, binocular refractive methods would limit accommodative stimulation and thus visual fatigue. However, these methods are little used in favour of conventional methods. It is therefore necessary to evaluate the interest of binocular refraction for the adjustment of night vision binoculars.

The purpose of this study is to compare refraction measurements by procedure in adult subjects free of ophthalmological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 ;
* Non-presbyopic subject;
* Stereoscopic acuity ≤ 60 arc seconds.

Exclusion Criteria:

* Accommodative insufficiency;
* Accommodative inertia;
* Compensation by orthokeratology (i.e. night lenses);
* Present or past binocular pathology (strabismus or amblyopia);
* Pregnant or nursing woman;
* Incomprehension of French (written and spoken).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Maximum convex equivalent sphere values | At visit 1 (day 1)
  Maximum convex equivalent sphere values obtained by the different refraction procedures under study.

SECONDARY OUTCOMES:
High contrast monocular acuity values | At visit 1 (day 1)
  High contrast monocular acuity values obtained by the different refraction procedures.
Low contrast monocular acuity values | At visit 1 (day 1)
  Low contrast monocular acuity values obtained by the different refraction procedures.
High contrast binocular acuity values | At visit 1 (day 1)
  High contrast binocular acuity values obtained by the different refraction procedures.
Low contrast binocular acuity values | At visit 1 (day 1)
  Low contrast binocular acuity values obtained by the different refraction procedures.
Difference between binocular perceptual assessment scores before and after subjective adjustment | Difference between visit 1 (day 1) and visit 2
  Difference between binocular perceptual assessment scores obtained by the different refractive procedures before and after subjective adjustment.
  Binocular perceptual assessment score will be obtained using visual analogue faces. The score will range from "excellent comfort" to "unbearable".

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided